CLINICAL TRIAL: NCT03573583
Title: Time Course Adaptations Using Deuterated Creatine (D3Cr) Method: A Pilot Study
Brief Title: Time Course Adaptations Using Deuterated Creatine (D3Cr) Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB201801249 - N; P30AG028740 (NIH)
Record Dates: First submitted 2018-06-05; First posted 2018-06-29 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Sarcopenia
Keywords: muscle mass; muscle loss; Deuterated creatine (D3Cr) dilution; older adults; resistance training; physical function
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The pilot study will be single-blind, parallel group, randomized controlled trial of 24 moderate to low functioning participants randomized in a 1:1 allocation ratio to a high-intensity Resistance Training group (RT) or a Successful Aging Health Education comparator group (HE) for 14 weeks.
Who Masked: Outcomes Assessor
Masking Description: To ensure concealment of the allocation, the randomization procedures will be performed by an investigator who are not involved in the assessments.
  The team assessing study outcomes will be masked to intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Training group (RT) (Experimental): The resistance training intervention will include a full body, resistance training performed three days per week.The intensity, volume, tempo, and progression will be based on the Federal Physical Activity guidelines
  Interventions: Behavioral: Resistance Training
- Successful Aging (Active Comparator): The comparator group will meet for stretching and health education classes every 2-5 weeks up to 7 total visits.
  Interventions: Behavioral: Successful Aging

INTERVENTIONS:
Behavioral: Resistance Training — The intensity, volume, tempo, and progression will be based on the Federal Physical Activity guidelines. The resistance training exercises will include mainly multi-joint exercises using selectorized machines. Each session will include upper body exercises (Chest Press, Shoulder Press, Seated Rows, Bicep curls, and Tricep Extensions) and lower body exercises (Leg Press, Leg Extension and Leg Curls, and Calf raise) that will be tailored to the participant needs.
  Other Names: RT; Strength Training; Weight Training
  Arms: Resistance Training group (RT)
Behavioral: Successful Aging — The successful aging will attend stretching and health lectures as a group . The topics might include, medication management, disease management (e.g. blood pressure, diabetes, arthritis, dementia, pain management, diet) and other health related matters.
  Other Names: HE; Health Education
  Arms: Successful Aging

SUMMARY:
The pilot study is to assess the feasibility of using a new method to measure muscle mass called Deuterated Creatine (D3Cr) method and thereby understand the role of muscle mass on functional outcomes in older adults.

DETAILED DESCRIPTION:
Muscle loss with age is considered to be an important cause of disability in older adults. However, current tools frequently used and recommended to measure muscle mass in trials have limitations: For example, DEXA (Dual-energy X-ray absorptiometry) and BIA (Bioelectrical impedance analysis)- both widely used in clinical trials cannot distinguish muscle tissue from non-muscle elements such as subcutaneous and intramuscular fat, skin, water and connective tissue.

Deuterated creatine (D3Cr) dilution is a novel promising method that provides an accurate measure of the functional contractile tissue, without including the non-contractile elements, by measuring total body creatine. Our preliminary cross-sectional results in men aged >65 years show functional muscle mass (FMM) assessed by D3-Cr to be significantly associated with performance outcomes and long-term outcomes, while DEXA showed no associations. However, these are observational data and cannot determine a causative role of muscle per se on functional outcomes.

Hence, the objective of the pilot study is to assess the feasibility of our proposed future study to evaluate the role of muscle mass on functional outcomes. Specifically, the pilot study will randomize moderate to low-functioning older adults to a resistance training program or successful aging health education program to assess recruitment yields, participant adherence, retention, training program design aspects, sample size, and the cost of the main trial. Further, the impact of these changes in FMM on short-term performance outcomes, such as strength, walking speed, SPPB, self-reported measures, and balance will be examined.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 70 or greater
* at high risk for mobility disability based on lower extremity functional limitations measured by Short Physical Performance battery (SPPB) with a score ≤ 8 out of 12
* could safely participate in the resistance training intervention as determined by medical history and physical examination.
* willing to give informed consent to be randomized to either the resistance training group or successful aging heath education comparison group and willing to follow the study protocol

Exclusion Criteria:

* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Myocardial infarction, major heart surgery, stroke, deep vein thrombosis, or pulmonary embolus in the past 6 months
* Lung disease requiring either oral or injected steroids, or the use of supplemental oxygen
* Short, portable mental status questionnaire with 3 or more errors
* Severe arthritis (either osteoarthritis or rheumatoid arthritis) that severely limits mobility
* Severe lower back or shoulder pain that can worsen with weight lifting exercises.
* Cancer requiring treatment in the past 1 year (Melanomas excluded)
* Any present or recent history of severe psychiatric illness including depression that might preclude providing informed consent, safe participation, or compliance (self-report and investigator judgement
* Development of chest pain or severe shortness of breath on the 400 m self-paced walk test
* Parkinson's disease or other serious neurological disorders; renal disease requiring dialysis; other illness of such severity that life expectancy is considered to be less than 12 months
* Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* Current consumption of more than 14 alcoholic drinks per week
* Uncontrolled hypertension (systolic blood pressure > 200 mm Hg and/or diastolic blood pressure >110 mm Hg)
* Currently on testosterone, Dehydroepiandrosterone (DHEA), or anabolic steroids.
* Undergoing physical therapy involving the lower extremities
* Currently enrolled in another randomized trial involving a pharmaceutical or lifestyle intervention. Observational studies are permitted
* Participation in progressive resistance exercise regimen ( ≥1 day/week) within the previous 6 months prior to screening.
* Weight change (intentional or not) over the last 6 months of > 5% of body or plan to lose or gain weight during the study
* Any other cardiovascular, pulmonary, orthopedic, neurologic, or other conditions that in the opinion of the local clinician would preclude participation and successful completion of the protocol

Temporary Exclusion Criteria:

* Recent bacterial/viral infection (e.g. pneumonia) (< 2 weeks);
* Acute febrile illness in past 2 months;
* Severe hypertension, e.g., SBP > 200 mm Hg, DBP > 110 mm Hg
* Major surgery or fracture or hip/knee replacement (< 6 months);
* Hospitalization within the last 6 months ( Not ER visits)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Manini, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health at the University of Florida, Gainesville, Florida
  - UF Institute on Aging Clinical and Translational Research Building, Gainesville, Florida

REFERENCES:
- [Result] Balachandran AT, Evans WJ, Cawthon PM, Wang Y, Shankaran M, Hellerstein MK, Qiu P, Manini T. Comparing D3-Creatine Dilution and Dual-Energy X-ray Absorptiometry Muscle Mass Responses to Strength Training in Low-Functioning Older Adults. J Gerontol A Biol Sci Med Sci. 2023 Aug 27;78(9):1591-1596. doi: 10.1093/gerona/glad047. PMID 36752568

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community using flyers, posters, and mass mailings. The eligibility criteria included men and women aged 70 years or older, who were at high risk for mobility disability based on lower extremity functional limitations measured by the Short Physical Performance Battery (SPPB) with a score of 9 or lower out of 12, and not participating in a structured exercise program, and not using strength exercises in the past 6 months.
Pre-assignment Details: A total of 54 participants were assessed for eligibilty and 33 were excluded ( 23 not meeting inclusion criteria (18 SPPB out of range) and 10 withdrew pre-randomization). Twenty-one participants met eligibility criteria and were subsequently randomized into 2 groups
Groups:
- Resistance Training Group (RT): The resistance training intervention will include a full body, resistance training performed three days per week.
  The intensity, volume, tempo, and progression will be based on the Federal Physical Activity guidelines
  Resistance Training: The intensity, volume, tempo, and progression will be based on the Federal Physical Activity guidelines. The resistance training exercises will include mainly multi-joint exercises using selectorized machines. Each session will include upper body exercises (Chest Press, Shoulder Press, Seated Rows, Bicep curls, and Tricep Extensions) and lower body exercises (Leg Press, Leg Extension and Leg Curls, and Calf raise) that will be tailored to the participant needs.
Period: Overall Study
Arm/Group | Resistance Training Group (RT) | Successful Aging
Started | 10 | 11
Completed | 8 | 10
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resistance Training Group (RT) | Successful Aging | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.4 (5.8) | 83.6 (5.4) | 82 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Short Physical Performance Battery Score [Mean (Standard Deviation); unit: units on a scale] — Short Physical Performance Battery Score (SPPB) is a measure of lower body physical performance consisting of three tests: a 4-meter usual gait speed test, five repeated chair stands, and three standing balance tests (side-by-side stance, modified tandem stance, tandem stance). Each component is scored from 0 to 4, with a total possible score ranging from 0 (worst performance) to 12 (best performance) by summing the individual scores.
  units on a scale | 6.7 (0.8) | 6.9 (1.6) | 6.8 (1.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2.] | 30 (3.3) | 30 (3.3) | 30 (3.3)
D3Cr Muscle Mass [Mean (Standard Deviation); unit: Kg] | 17.3 (4.2) | 18 (4.9) | 17.65 (4.6)
DXA Appendicular Lean Mass [Mean (Standard Deviation); unit: kg] | 16.4 (4.2) | 17.6 (4.6) | 17 (4.4)
DXA Lean Body Mass [Mean (Standard Deviation); unit: Kg] | 44.2 (11.3) | 42.2 (8.9) | 43.2 (10.1)
DXA Fat Mass [Mean (Standard Deviation); unit: Kg] | 35.8 (8.3) | 34.4 (5.2) | 35.1 (6.75)
Number of Participants with College Education or Higher [Count of Participants; unit: Participants] | 9 | 10 | 19
Number of Participants taking Medications for High Blood Pressure [Count of Participants; unit: Participants] | 5 | 8 | 13
Number of Participants taking Medications for Diabetes [Count of Participants; unit: Participants] | 0 | 3 | 3
Number of Participants taking Medications for High Cholesterol [Count of Participants; unit: Participants] — Number of participants taking medications for managing high cholesterol assessed via self-reports.
  Participants | 5 | 3 | 8
Number of Partcipants who had Cancer. [Count of Participants; unit: Participants] — Number of participants who had cancer, a malignant growth or tumor (excluding uterine fibroids and minor skin cancer) requiring treatment in the last year.
  Participants | 1 | 0 | 1
Number of participants with Lung Disease [Count of Participants; unit: Participants] — Number of participants that have chronic lung disease such as chronic bronchitis, COPD, asthma, or emphysema that was diagnozed by a doctor.
  Participants | 0 | 3 | 3
Number of Partcipants who had a Stroke [Count of Participants; unit: Participants] — Number of partciants had a stroke or brain hemorrhage as diagnozed by a doctor and had to be hospitalized?
  Participants | 1 | 0 | 1
Number of Partcipants who had Myocardial Infarction or Major Heart Surgery [Count of Participants; unit: Participants] — Number of participants who had a heart attack, major heart surgery, stroke, deep vein thrombosis, or pulmonary embolus in the past 6 months
  Participants | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Muscle Mass
Description: Change in Muscle mass measured using D3Cr
Time Frame: Baseline and week 16
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Resistance Training Group (RT) | Successful Aging
Number analyzed (Participants) | 10 | 11
Kg | 3.47 (2.01) | 1.19 (1.70)
Statistical Analysis 1: Comparison: Resistance Training Group (RT) vs Successful Aging; Continuous variables were expressed as mean (SD) and categorical variables were as frequencies and percentages. A 2-sided independent-sample t test was used to compare group differences in change scores. Change scores were calculated as Week 16 measurements minus baseline measurements. Statistical analyses were done by a blinded statistician without knowledge of group membership; Test type: Superiority; p = 0.03, ANCOVA — No formal adjustment for type I error due to the pilot nature of the study. All significance tests were 2-tailed and an alpha level of 0.05 was required for significance; Adjusted for baseline score; Mean Difference (Final Values) = 2.29, 95% CI 2-sided [0.22 to 4.36]

2. Secondary Outcome: Appendicular Lean Mass (ALM)
Description: Change in ALM by dual-energy x-ray absorptiometry (DEXA)
Time Frame: Baseline and week 16
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Resistance Training Group (RT) | Successful Aging
Number analyzed (Participants) | 10 | 11
Kg | 0.81 (0.68) | -0.23 (0.70)
Statistical Analysis 1: Comparison: Resistance Training Group (RT) vs Successful Aging; Test type: Superiority; p = 0.009, ANCOVA; Adjusted for baseline score; Mean Difference (Final Values) = 1.04, 95% CI 2-sided [0.31 to 1.77]

3. Secondary Outcome: Lean Body Mass (LBM)
Description: Change in LBM assessed using DXA
Time Frame: Baseline, and Week 16
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Resistance Training Group (RT) | Successful Aging
Number analyzed (Participants) | 10 | 11
Kg | 1.10 (1.44) | -0.19 (0.93)
Statistical Analysis 1: Comparison: Resistance Training Group (RT) vs Successful Aging; Test type: Superiority; p = 0.07, ANCOVA; Baseline as covariate; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [-0.10 to 2.67]

4. Secondary Outcome: Correlation Between Changes in Muscle Mass
Description: Correlation between longitudinal changes in D3 Cr muscle mass (MM) and DXA appendicular lean mass (ALM)
Time Frame: Baseline and Week 15
Population: We want to analyze the correlation between DXA ALM and D3Cr muscle mass. Hence, the two groups are combined to calculate the correlation of DXA ALM compared to D3Cr muscle mass in all the participants rather than individual groups.
Measure: Mean (95% Confidence Interval); unit: Pearson Correlation Coefficient
Groups:
- Total Participants: Combined both groups (Successful Aging + Resistance training) into one group.
Arm/Group | Total Participants
Number analyzed (Participants) | 18
Pearson Correlation Coefficient | 0.19 [-0.35 to 0.64]
Statistical Analysis 1: Comparison: Total Participants; Test type: Other — Pearson's correlation coefficients, along with their 95% confidence intervals (CIs); p = 0.49, Pearson's Correlation coefficient; Pearson's Correlation coefficient = 0.19, 95% CI 2-sided [-0.35 to 0.64]

ADVERSE EVENTS:
Time Frame: 15 weeks
Arm/Group | Resistance Training Group (RT) | Successful Aging
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

LIMITATIONS AND CAVEATS:
Our study has several limitations. First, the sample size was relatively small. Clearly, the study needs to be replicated with a larger sample to make definitive statements. Although it is considered a strength in some respects, the results are only applicable to low-functioning older adults. Additional measures of body composition were not included, but would have allowed additional comparisons (eg, whole-body MRI or a 4-compartment model) with D3Cr.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT03573583/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT03573583/ICF_001.pdf